CLINICAL TRIAL: NCT01606163
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Multiple-dose, Dose Escalation Study to Assess the Safety and Pharmacokinetics of GC1102 (Hepabig-Gene) in Healthy Male Adults
Brief Title: Safety and Pharmacokinetics Study of Healthy Male Adults When Repeatedly Administered Through Intravenous Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GC1102
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- group 1 (Experimental): 1. Drug:GC1102
  2. Amount:3ml (30,000IU)
  Interventions: Biological: GC1102
- group 2 (Experimental): 1. Drug: GC1102
  2. Amount: 5ml(50,000IU)
  Interventions: Biological: GC1102
- group 3 (Experimental): 1. Drug: GC1102
  2. Amount: 8ml (80,000IU)
  Interventions: Biological: GC1102
- group 4 (Placebo Comparator): drug: JW normal saline
  Interventions: Other: JW normal saline

INTERVENTIONS:
Biological: GC1102 — 1. Description: GC1102 IV bolus injection during 10~ 30 seconds.
  2. Amount: group1-3ml, group2-5ml, group3-8ml
  3. Subject number: group1-8, group2-8, group3-8
  4. Administration time: 1day, 2day, 3day, 4day, 5day, 6day, 7day(total: 7 times)
  Other Names: Hepabig_Gene
  Arms: group 1; group 2; group 3
Other: JW normal saline — 1. Description: Normal saline IV bolus injection through 10~ 30 seconds.
     * Each 3 subjects of this placebo comparator group will match with group 1,2,3 respectively. Placebo comparator subjects in each group will be treated with same condition of each group(group 1, group 2, group 3) except being administered JW normal saline.
  2. Subject number: 9
  3. Administration time: 1day, 2day, 3day, 4day, 5day, 6day, 7day(total: 7 times)
  Other Names: saline solution
  Arms: group 4

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics of healthy male adults when subjects are repeatedly administered GC1102 (Hepabig_Gene) through intravenous injection.

ELIGIBILITY:
Inclusion Criteria:

* Those who are healthy, male adult aged 20 years- 45 years when screened.
* Those whose body weights are over 45kg when screened, and whose BMI scores are 19kg/㎡-28 kg/㎡.
* Those whose HBs-Ag, HBc-Ab(IgM), HBc-Ab(IgG), HBV DNA quantitative are all negative when screened.
* Those whose HBs-Ab(titer) in blood is below 500 IU/L when screened.
* Those who agree to use double protective contraceptive measures from one days before administration of first investigative drug to last follow-up visit(protective contraceptive measures using more than 2 ways among a male condom, a female condom of sex partner, a spermicide of sex partner, an intrauterine device(IUD) of sex partner, a diaphragm of sex partner and a cervical cap of sex partner), and not to provide sperm.
* Those who voluntarily decide to follow matters that require attention of this study and give written consent to participate in this clinical trial.
* Those who can visit the medical center to be monitored, and agree to collect blood during study period.

Exclusion Criteria:

* Those who have GC1102 anti-body when screened
* Those who have a clinically meaningful disease or history concerning liver, kidney, alimentary system, respiratory system, musculoskeletal system, endocrine system, neuropsychiatry system, blood tumor system, cardiovascular system.
* Those who have anaphylaxis of drug allergy including HBIG or who have allergy disease requiring treatment.
* Those who have immunodeficiency disease now.
* Those who have an anamnesis of Guillain-Barre syndrome.
* Hemophiliac patients who have a risk of serious bleeding when getting a shot through intravascular injection or those who are being administered anticoagulants
* Those who are administered live vaccine parenterally within 120 days from being administered first investigative drug. (ex: measles vaccine, epidemic parotitis vaccine, rubella vaccine, cholera vaccine, chickenpox vaccine)
* Those who are administered interferon or antiviral agents within 120 days from being administered first investigative drug. (except for topical medication)
* Those who showed signs of an acute fever(over 38℃) within 72 hours from being administered first investigative drug.
* Those who showed signs of acute disease within 14 days from being administered first investigative drug.
* Those who donated whole blood within 60 days or ingredient blood within 30 days from being administered first investigative drug or those who are administered blood transfusion within 30 days from being administered first investigative drug.
* Those who took other investigative drugs within 60 days from being administered first investigative drug.
* Those who took herbal medicine within 30 days from being administered first investigative drug or took ethical drug(ETC) within 14 days or took over-the- counter drug(OTC) within 7 days from being administered first investigative drug.(but, Those who meet other conditions can join the clinical trials according to investigator's decision)
* Those who drink excessively caffeine-contained beverage, excessive alcohol, and who are smokers( caffeine> 5 units/ day, alcohol>21 units/ week, cigarette> 10 pieces) or have a history of alcoholism
* Those who have a history of drug addiction, or showed positive response of urine-drug screening examination (ex: amphetamine, methamphetamine, barbiturate, cocaine, opiate, benzodiazepines, cannabinoid, methadone, etc)
* Those who showed positive sign of serum test(A-type hepatitis test(HAV IgM Ab), C-type hepatitis test(HCV Ab screening), HIV test(HIV Ag & Ab), Syphilis high quality reagin test.
* Those whose serum creatinine, ALT, AST, or total bilirubin exceeded the standard 1.5 times by the diagnostic lab test.
* Those who cannot eat standard meals provided by Seoul Asan medical center.
* Those who are judged disqualified to join clinical trials by investigator for other causes.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Safety of GC1102 when repeatedly administered by intravenous injection to healthy male adults | screening, -1d, 1d, 2d, 3d, 4d, 5d, 6d, 7d, 8d, 9d, 14d, 21d, 28d
  * Adverse event
  * Diagnostic examinations
  * Physical examinations
  * Vital signs
  * ECG(electrocardiogram)
  * Check of concomitant drug

SECONDARY OUTCOMES:
Pharmacokinetics of GC1102 when repeatedly administered by intravenous injection to healthy male adults | 1)1d:predose(0h), 0.5, 1, 2, 5, 9, 14 hours after dose 2) 2d~6d:predose(0h) 3) 7d:predose(0h), 0.5, 1, 2, 5, 9, 14 hours after dose 4) 8d, 9d, 14d, 21d, 28d: 0h
  * Terminal elimination half-life (t½β)
  * Maximum and Average concentration at steady state(Cmax,ss, Cav,ss,)
  * Area-under the concentration-time curve within a dosing interval at steady state (AUCτ,ss)
  * Clearance (CL)
  * Volume of distribution at steady state (Vd,ss)
  * Mean residence time (MRT)
  * Accumulation Index (AI)

CONTACTS AND LOCATIONS:
Overall Officials: Kyun-Seop Bae, MD, PhD, Principal Investigator — Department of clinical pharmacology and therapeutics
Locations (1):
- Department of clinical pharmacology and therapeutics, Seoul, South Korea